CLINICAL TRIAL: NCT06893705
Title: Effects OF Pilates Exercises on Pain, Functional Disability and ROM Among School Going Children With Text Neck Syndrome
Brief Title: Pilates Exercises on Pain, Functional Disability and ROM Among Children With Text Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/24/0745
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Children, Adult
Keywords: Pilates; Neck Pain; Range of Motion; School Children; Text Neck
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial performed through convenient sampling, in which 24 TNS children with the age 12-17 years will be taken randomly after screening and meeting inclusion criteria. Children will be divided in two groups. Control Group will receive conventional therapy for 50 min in a day for 3 days per week. Experimental Group will receive Pilates with Conventional Therapy for 50 min in a day for 3 days per week. Pre values were taken at 1st week , 3rd week and post values of intervention will be taken after 6th week to measure the effects of both therapies.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Control : For group A Conventional Therapy Program for 50 min, 3 days per week during a 6 week period.
  Interventions: Other: Conventional Therapy
- Group B (Experimental): Experimental: For group B 25 min of pilates and 25 min of conventional therapy 3 days per week during a 6 week period
  Interventions: Other: Pilates+Conventional Therapy

INTERVENTIONS:
Other: Conventional Therapy — Conventional Therapy Group: Group A will be control group which will receive conventional physical therapy program for the affected neck like stretching exercises, active range of motion exercise, and neck isometrics for 6 weeks (3 sessions per week).
  Arms: Group A
Other: Pilates+Conventional Therapy — Group B will be experimental group, which will receive Pilate's exercises like cat stretch, swan dive/roll up along with conventional therapy for 6 weeks(3 sessions per week). In each session there will be 25 minutes of conventional therapy and 25 minutes of Pilate's exercises program.
  Arms: Group B

SUMMARY:
Text Neck' is a term used to describe a posture that is caused by leaning forward for long period of time such as reading or texting on smartphone. Neck pain, discomfort, reduced function and limited range of motion are the signs of text neck. Forward head posture is the most common cervical issue in the sagittal plane. Neck pain interferes with daily life activities. Pilates exercise program is the most appropriate exercise program for the prevention of forward head posture. For improvement with neck pain and activity limitation 24 Children with age 12-17 year will be randomly assign in 2 groups.

Group A will receive conventional physical therapy program for the affected neck like stretching exercises, active range of motion exercise, and neck isometrics for 6 weeks (3 sessions per week). The treatment duration will be of 50 min. On the other hand Group B will receive Pilate's exercises like cat stretch, swan dive/roll up along with conventional therapy for 6 weeks(3 sessions per week). In each session there will be 25 minutes of conventional therapy and 25 minutes of Pilate's exercises program. Then evaluate both groups on follow up.

All data will be collected from Gov. High School Niaz Baig by using Visual Analogue Scale, Functional Disability Index questionnaire and Goniometer. The reliability and validity of tools are mentioned.

The duration of study will be 6 months. Data will be analyzed with the help of SPSS 25.

DETAILED DESCRIPTION:
Text Neck' is a term used to describe a posture that is caused by leaning forward for long period of time such as reading or texting on smartphone. Neck pain, discomfort, reduced function and limited range of motion are the signs of text neck. Forward head posture is the most common cervical issue in the sagittal plane. Neck pain interferes with daily life activities. Pilates exercise program is the most appropriate exercise program for the prevention of forward head posture. It focuses on postural alignment, which results in increasing craniovertebral angle and decreasing pain. Improving text neck is very important because it can enhance an individual's ability to perform everyday activities.

A randomized controlled trial will be conducted through convenient sampling. Data will be collected from Allied school and The Trust School, Lahore. Sample size of 24 subjects, with age group between 12 to 17 years will be taken. Data will collected from participants that use smart phone for more than 4hr/day. Participants with cervical fracture, trauma and scoliosis will be excluded. Outcome measure will be taken using Visual Analogue Scale (VAS) for pain, Functional Disability Inventory (FDI) for function and Universal Goniometer (UG) for range of motion. An informed consent will be taken. Subjects will be randomly allocated into two groups: experimental group will receive Pilates exercise program like cat/chest stretch, swan dive/spine twist in addition to designed conventional therapy, while the control group will receive designed conventional therapy for the affected neck like stretching exercises, neck isometrics and active range of motion exercises. The treatment duration will be of 6 weeks and 50min/day. Data will be analyzed on SPSS version 25; the normality of the data will be checked and tests will be applied according to the normality of the data either it will be a parametric or non-parametric test based on the normality.

ELIGIBILITY:
Inclusion Criteria:

* CVA < 48 degree
* Age 12 to 17 years
* Both male and female
* Mobile phone usage more than 4 hr. /day
* More than one year of using any electronic gadgets.

Exclusion Criteria:

* Vertigo
* Kyphosis
* Scoliosis
* Trauma/Cervical Fracture
* Torticollis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
FDI(Functional Disability Inventory Questionnaire) | Baseline,3rd week, 6th week
  The functional disability inventory: measures a neglected dimension of child health status. It assesses activity limitations in children and adolescents. High score indicate 'greater functional disability'. A clinical tool for measuring impact of neck pain on patient's daily life. It consists of 15 items. Internal consistency reliability is excellent(R=0.86 to 0.91)(p<0.05)
VAS(Visual Analogue Scale) | Baseline, 3rd week,6th week
  A clinical tool used for measuring the intensity of pain. It is a horizontal 10cm line with '0' at one end which indicate no' pain', and '1' at the other end which indicate 'worst pain'. Subject is asked to mark his/her pain according to the severity.(R=0.97)(p=0.02)
Goniometer | Baseline,3rd week, 6th week
  Goniometer is used to measure range of motion .It also measures cervical ROM in flexion, extension, rotation and side bending. Reliability score of cervical goniometer ranged from(R= 0.999 to 0.931) (p<0.05) for cervical region

CONTACTS AND LOCATIONS:
Overall Officials: Aira Eman, MS-PPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Muhammad Asif Javed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] David D, Giannini C, Chiarelli F, Mohn A. Text Neck Syndrome in Children and Adolescents. Int J Environ Res Public Health. 2021 Feb 7;18(4):1565. doi: 10.3390/ijerph18041565. PMID 33562204